CLINICAL TRIAL: NCT02971969
Title: A Long-Term Follow-up Study to Evaluate the Safety, Tolerability, and Efficacy of Adeno-Associated Virus (AAV) rh10-Mediated Gene Transfer of Human Factor IX in Adults With Moderate/Severe to Severe Hemophilia B
Brief Title: Long-Term Safety, Tolerability, and Efficacy of DTX101 (AAVrh10FIX) in Adults With Moderate/Severe to Severe Hemophilia B
Status: Completed | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 101HEMB02; 2016-003430-25 (EudraCT Number)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Hemophilia B
Keywords: gene therapy; Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
A long-term follow-up study to evaluate the safety, tolerability, and efficacy of DTX101 in adult males with moderate/severe to severe hemophilia B.

DETAILED DESCRIPTION:
Hemophilia B is an X-linked recessive genetic bleeding disorder caused by mutations in the factor IX (FIX) gene. FIX is produced in the liver and is critical for fibrin clot formation. Hemophilia B is characterized by frequent, spontaneous internal bleeding that can lead to chronic arthropathy (joint damage), intracranial hemorrhage, and even death. In patients with moderate/severe to severe hemophilia B, the majority of bleeding episodes occur in the joints and, if not treated, lead to debilitating damage and a decreased quality of life.

Study 101HEMB02 is a long-term follow-up study to evaluate the safety, tolerability, and efficacy of AAVrh10-mediated gene therapy of human FIX in subjects with moderate/severe to severe hemophilia B. The primary objective of the study is to determine the long-term safety and efficacy of DTX101 following a single IV infusion (administered during Study 101HEMB01) in adults with moderate/severe to severe hemophilia B.

This study was previously posted by Dimension Therapeutics, which has been acquired by Ultragenyx.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Completed the Week 52 visit in Study 101HEMB01.
3. Willing to stop prophylactic treatment with recombinant FIX at specified time points during the study if medically acceptable.
4. Willing, able, and committed to comply with scheduled study site visits, study procedures, and requirements.

Exclusion Criteria:

1. Planned or current participation in another interventional clinical study that may confound the efficacy or safety evaluation of DTX101 during the duration of this study.
2. Any clinically significant medical condition that, in the opinion of the investigator, would pose a risk to subject safety or would impede the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males with moderate/severe to severe Hemophilia B previously enrolled in 101HEMB01 clinical study
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-01; Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events by dosing group | 208 weeks
Change from baseline in FIX activity level | 208 weeks

SECONDARY OUTCOMES:
Number of bleeding episodes requiring recombinant FIX infusion | 208 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (5):
- United States (3):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UF CRC - Clinical Research Center, Gainesville, Florida
  - University of Michigan Hospital and Health Systems, Ann Arbor, Michigan
- United Kingdom (2):
  - Haemophilia, Haemostasis & Thrombosis Centre, Basingstoke, Hampshire
  - Manchester Haemophilia Comprehensive Care Center, Manchester

REFERENCES:
- [Derived] Pipe S, Poma A, Rajasekhar A, Everington T, Sankoh S, Allen J, Cataldo J, Crombez E. Gene therapy for hemophilia B: results from the phase 1/2 101HEMB01/02 studies. Blood Adv. 2025 Jun 24;9(12):2980-2987. doi: 10.1182/bloodadvances.2024015184. PMID 40197980